CLINICAL TRIAL: NCT02003651
Title: Efficacy of Ingesting Gaia Herb's Quick Defense Product in Reducing Acute Respiratory Illness Symptomatology in Women: a 12-Week, Double Blind, Placebo-Controlled Randomized Trial
Brief Title: Echinacea and Acute Respiratory Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Gaia Herbs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0064
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2015-01

CONDITIONS: Acute Respiratory Infections
Keywords: Common cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quick Defense (Experimental): 250 mg E. purpurea root and 83 mg E.angustifolia root standardized to 10 mg alkylamides, and 210 mg of a proprietary synergistic extract blend containing andrographis paniculata leaf, black elderberry berries, sambucus nigra, ginger root, and zingiber officinale
  Interventions: Dietary Supplement: Quick Defense
- Placebo (Placebo Comparator): Placebo will contain the excipients vegetable glycerin and olive oil. Placebo and echinacea capsules will be colored green and contain the same proportions of inert ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Quick Defense — Echinacea product from Gaia Herbs.
  Arms: Quick Defense
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of ingesting an alkylamide-rich echinacea root product (Quick Defense, Gaia Herbs) for 2 days immediately following each onset of acute respiratory illness (ARI) symptomatology during a 12-week period in the winter and early spring in women.

Hypothesis: Subjects randomized to Quick Defense compared to placebo over a 12-week period will experience reduced ARI symptomatology, both acutely during each ARI episode and collectively over the entire 12-week study period.

DETAILED DESCRIPTION:
The common cold is an acute respiratory illness (ARI) and the most frequent illness people experience, with economic costs estimated at $40 billion per year (Ann Intern Med 2010;153:769-777). Hundreds of different types of viruses cause the common cold, and etiologic agents include rhinovirus, coronavirus, influenza, parainfluenza, respiratory syncytial virus, adenovirus, enterovirus, and metapneumovirus.

The purple coneflower (E. angustifolia and E. purpurea) is one of the most popular herbal supplements in North America and Europe. Echinacea preparations are marketed to provide protection and treatment for the common cold. Reviews and meta-analyses provide modest support for the use of Echinacea in the prevention and treatment of the common cold (Can Fam Physician 2011;57:31-6; Cochrane Database Syst Rev 2006 Jan 25;(1):CD000530; Lancet Infect Dis 2007;7:473-80; Clin Ther. 2006 Feb;28(2):174-83). One meta-analysis concluded that echinacea decreased the odds of developing the common cold by 58% and the duration of a cold by 1.4 days (Lancet Infect Dis 2007;7:473-80).

Echinacea products vary in their composition, due to the use of different species, plant parts, extraction methods, and addition of other components (Planta Med 2008;74:633-7). Some preparations are based on the stabilized fresh juice of aerial parts of E. purpurea, and are rich in hydrophilic derivatives such as polysaccharides and glycoproteins. Other echinacea products come from an extract of root material and contain more lipophilic compounds including N-alkylamides (Ann Intern Med 2010;153:769-777).

Studies indicate that echinacea preparations containing N-alkylamides are bioavailable in humans and can suppress stress-related cellular immune responses (Life Sci 2009;85(3-4):97-106). Echinacea preparations containing N-alkylamides have been linked to multiple immune-modulatory activities including enhanced macrophage phagocytic activity and suppression of the proinflammatory responses of epithelial cells to viruses and bacteria (J Biomed Biotechnol. 2012;2012:769896). Echinacea preparations appear to have low potential to generate cytochrome P450 (CYP 450) drug-herb interactions, and there are no verifiable reports of drug-herb interactions. The estimated risk of taking echinacea products is 1 in 100,000, and thus do not appear to pose a risk to consumers (Mol Nutr Food Res. 2008;52(7):789-98).

Barrett et al. (Ann Intern Med 2010;153:769-777) enrolled subjects within 36 hours of illness onset, and administered echinacea tablets (or placebo) containing 675 mg E. purpurea root standardized to 2.1 mg alkamides and 600 mg E. angustifolia root standardized to 2.1 mg alkamides. Subjects consumed two tablets at enrollment, followed by two-tablet doses three more times within 24 hours of enrollment. Dosing then went to one tablet four times daily for the next four days. Thus, each participant ingested the equivalent of 10.2 g of dried echinacea root during the first 24 hours and the equivalent of 5.1g during each of the next four days. Results were in the direction of benefit, amounting to an average half day reduction in the duration of a week-long cold, or an approximate 10% reduction in overall severity.

The proposed study will build upon the study by Barrett et al., (2010) by initiating 2-day use of an alkylamide-rich echinacea root product (Quick Defense, Gaia Herbs) within the first few hours of each ARI onset throughout a 12-week period in the winter/early spring.

1. DESIGN GUIDELINES:

   1. Following recruitment, subjects will come to the ASU-NCRC Human Performance Lab (visit 1 or pre-study visit) for orientation and to provide voluntary consent to join the study. All subject inclusion and exclusion criteria must be maintained during the study.
   2. Subjects will fill in a medical health questionnaire to verify medical history and lifestyle habits (completed and handed in at visit 1).
   3. Subjects will have two additional laboratory visits (6-weeks and 12-weeks) at the ASU-NCRC Human Performance Laboratory.

      At each of the three lab visits, body weight and percent body fat (Tanita BIA scale) will be measured. Height will be measured at the pre-study visit. At each lab visit, subjects will also record responses to 6-week retrospective symptom logs. At the pre-study and 6-week study visits, subjects will be given 6-week daily log books, the Wisconsin Upper Respiratory Symptom Survey (WURSS-24), to assess symptoms related to the common cold. Subjects will turn this in during the 6-week and 12-week visits. Subjects will fill in a 6-week retrospective WURSS-24 during visit 1. Subjects will be interviewed by the lab staff at weeks 6 and 12 to determine whether there have been any changes in their medical history or medication use.
   4. Subjects (N=40-46) will be randomized to Quick Defense or placebo groups for 12 weeks (thus two independent groups with 20-23 subjects). Supplements will be administered in a double-blinded manner, with the code held by Gaia Herbs until the end of the study.
2. SUPPLEMENT:

Echinacea (Quick Defense) and identical placebo capsules will be manufactured by Gaia Herbs (Brevard, NC). Gaia Herbs will conduct an analysis of their product to verify supplement content. Two echinacea capsules will contain the equivalent of 250 mg E. purpurea root and 83 mg E.angustifolia root standardized to 10 mg alkylamides, and 210 mg of a proprietary synergistic extract blend containing andrographis paniculata leaf, black elderberry berries, sambucus nigra, ginger root, and zingiber officinale (see label above). Capsule excipients will include vegetable glycerin and olive oil, with the capsule containing vegetable cellulose. Placebo and echinacea capsules will be colored green and contain the same proportions of inert ingredients.

DOSING REGIMEN:

During the 12-week study, subjects will take 2 capsules 5 times daily (approximately every 3 hours) for 2 days each time they feel symptoms of an acute respiratory illness (ARI) are starting. Thus each subject will ingest the equivalent of 3.4 grams of dried echinacea root during the first two days of ARI onset. No additional echinacea (or placebo) capsules will be taken after the first two days of illness onset until the next ARI episode is experienced.

c. COMMON COLD SYMPTOMS: The Wisconsin Upper Respiratory Symptom Survey (WURSS-24) will be used to assess common cold illness severity and symptoms (see attached questionnaire). Scores from the WURSS-24 include: 1) Global severity score; 2) Symptom score; 3) Function ability score (Barrett et al., 2009). The WURSS-24 (short version to be used in this study) includes 10 items assessing symptoms (running nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion, feeling tired), 9 items assessing functional impairments (think clearly, sleep well, breathe easily, walk-climb stairs-exercise, accomplish daily activities, work outside the home, work inside the home, interact with others, live your personal life), and 1 item assessing global severity and global change. Subjects will fill in the one-page WURSS-24 at the end of each day during the 12-week monitoring period. This 12-week period will cover the winter and early spring period of 2014. From the responses recorded during the 84-day study, an ARI severity score will be calculated by summing the daily ARI global severity score (0=not sick, 1=very mild ARI to 7=severe). The ARI symptom score for the 84-day period will be calculated by summing all 10 symptom scores for each day's entry (0=do not have this symptom, 1=very mild to 7=severe). In similar fashion, the ARI function ability score for the 84-day period will be calculated by summing all 9 function scores for each day's entry (0=do not have this symptom, 1=very mild to 7=severe). Separate scores will be calculated comparing groups for each illness episode recorded by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult women, ages 18 to 55 years.
* Non-smokers.
* Willingness to avoid the use of antibiotics, antivirals, nasal steroids, decongestants, antihistamines, combination cold formulas, echinacea, zinc, or vitamin C during the 12-week study.
* Willingness to maintain normal dietary and physical activity patterns during the 12-week intervention, and not make formal attempts to lose body weight.

Exclusion Criteria:

* Current history of autoimmune or immune deficiency disease.
* History of moderate to severe allergic rhinitis with sneezing or itching of the nose or eyes during the winter/early spring.
* Current history of asthma with coughing, wheezing, or shortness of breath.
* Pregnant or planning to be pregnant during the study.
* History of gastrointestinal upsets, rashes, or allergic reactions to Echinacea.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Common cold symptoms | 12-weeks
  The Wisconsin Upper Respiratory Symptom Survey (WURSS-24) will be used to assess common cold illness severity and symptoms (see attached questionnaire). Subjects will fill in the one-page WURSS-24 at the end of each day during the 12-week monitoring period. This 12-week period will cover the winter and early spring period of 2014. From the responses recorded during the 84-day study, an ARI severity score will be calculated by summing the daily ARI global severity score (0=not sick, 1=very mild ARI to 7=severe). The ARI symptom score for the 84-day period will be calculated by summing all 10 symptom scores for each day's entry (0=do not have this symptom, 1=very mild to 7=severe). In similar fashion, the ARI function ability score for the 84-day period will be calculated by summing all 9 function scores for each day's entry (0=do not have this symptom, 1=very mild to 7=severe). Separate scores will be calculated comparing groups for each illness episode recorded by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- ASU-NCRC Human Performance Lab, Kannapolis, North Carolina, United States